CLINICAL TRIAL: NCT03300037
Title: HYpopnea and Apnea Detection and Treatment Performance of a New cardiOreSpiratory Holter Monitor
Acronym: HYPNOS
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: IAHO02
Record Dates: First submitted 2017-08-03; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Kinesthetic stimulation — The kinesthetic actuator is placed on the skin near the ear and emits vibrations.

SUMMARY:
The HYPNOS study is an acute feasibility study to validate a new device for automatic detection and treatment of sleep apnea syndrome. The system is known as the PASITHEA system and it will perform the following tasks:

* Detect apneas and hypopneas in real time, based on physiological signals acquired with a cardiorespiratory holter (nasal air flow, heart rate and blood oxygen saturation (SaO2))
* Upon detection of apnea or hypopnea events, trigger kinesthetic stimulation of mechanoreceptors of the skin close to the mastoid bone

The primary objective is to verify that the PASITHEA system is able to detect apneas and hypopneas reliably.

The main secondary objective of the study is to assess the effect of kinesthetic stimulation on reducing the number of sleep respiratory disorders.

Another objective of the study is to verify the safety of the PASITHEA system.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years.
* Patient with diagnosed severe obstructive sleep apnea syndrome (AHI > 30/h and > 80% of obstructive events diagnosed on polysomnography or polygraphy performed less than 6 months ago )
* Patient free from CPAP treatment or any other SAS treatment for at least 3 months
* Patient with stable psychotropic medication since the diagnostic polysomnography or polygraphy exam
* Patient has signed the informed consent

Exclusion Criteria:

* Patients sleeping less than 4 hours per night
* Patients suffering from respiratory failure or periodic breathing (cheynes stokes)
* Obese patient (BMI>40kg/m2)
* Diabetic patient with autonomic dysfunction
* Vulnerable patient in accordance with article L1121-6 of CSP
* Patient with progressive malignant pathology
* Patient already involved in another clinical study that could affect the result of this study
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe untreated obstructive SAS patients
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Performance of real-time detector of apnea and hypopnea: sensitivity and positive predictive value of the detector will be calculated when comparing automatically detected respiratory events to gold-standard PSG scoring of apnea/hypopnea events. | 1 night
  During the night of the recording, the PASITHEA system and the PSG will be positioned in parallel. PSG-scored events will be matched with the output of the real-time detector: a true positive event is defined as an event detected less than 10 seconds before or within the duration of a PSG-annotated events. Apneas detected as hypopneas (and reciprocally) will be regarded as true positives. Sensitivity and positive predictive value will be calculated as per conventional definintion and the 9% confidence interval will be calculated using the Wilson score.

SECONDARY OUTCOMES:
Safety: number of adverse events with treatment ON or OFF as defined by ISO 14155, rev 2011 | 1 night
  All adverse events will be recorded and assessed according to ISO 14155, rev 2011

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Angers, Angers
  - Laboratoire du sommeil et d'EFCR; Hopital Michallon, Grenoble
  - CHU Montpellier, Montpellier
  - CHU Rennes, Rennes
  - University Hospital Tours, Tours

IPD SHARING:
Plan to Share IPD: No